CLINICAL TRIAL: NCT05110456
Title: Starting Before Birth to Prevent Maternal Mental Health Problems: "Parents and Babies" Program (Programme "Toi, Moi, Bébé")
Brief Title: To Evaluate the Effectiveness of a Virtual and Telephone Intervention for the Prevention of Postpartum Depression in Women at Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Hewitt Foundation (Unknown)
Responsible Party: Principal Investigator, Sylvana M Côté, Researcher at the research center of the university hospital of saint justine, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-3210
Record Dates: First submitted 2021-10-13; First posted 2021-11-08 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to an online cognitive behavioural intervention without telephone support (No Intervention): The control group will receive a fully automated version of the virtual intervention without telephone support
- Cognitive-Behavioral Therapy (CBT) and interpersonal counseling with telephone support. (Experimental): The experimental group will receive an online cognitive behavioural intervention with weekly telephone support
  Interventions: Behavioral: Telephone support

INTERVENTIONS:
Behavioral: Telephone support — Participants will receive 10 telephone counseling calls by trained coaches: 9 during pregnancy (one call/week) and 1 at 6 weeks postpartum. We have included individual telephone calls by a trained coaches aimed to :
  1. encourage the use of online material;
  2. identify strategies for overcoming obstacles;
  3. help apply content to real-life settings; and
  4. underscore the participants' success in using effective coping strategies
  Arms: Cognitive-Behavioral Therapy (CBT) and interpersonal counseling with telephone support.

SUMMARY:
Women's perinatal mental health problems can create a cascade of short- and long-term negative influences for the mother, child, and the family as a whole. To prevent these impacts, preventive online and telephone interventions exist, but need to be tested and improved to develop this type of support to women in Quebec. The Parents & Babies program, which is a distance learning course, followed during pregnancy and accompanied by telephone follow-up, aims to improve the mental health of future parents.The investigators seek to evaluate the effect of the intervention of the Parents & Babies program offered with telephone support compared to the course offered without telephone follow-up.

DETAILED DESCRIPTION:
The Parents & Babies intervention to be evaluated is an adaptation of the existing, evidence-based Mothers & Babies program which has shown efficacy in four clinical trials for the prevention of postpartum depression through in-person (group or individual) counseling

The Parents & Babies program was adapted to be virtual and include: 1) specific modules for the mother-partner dyad; 2) third-wave cognitive behavioral therapy (CBT) strategies targeting well-being, relaxation, mindfulness, self-compassion, and gratitude; 3) confinement and social distancing related material. Participants follow the program online or with a paper workbook and are called weekly by a member of the intervention team.

Participants will fill out three questionnaires (online or by telephone) at 12-25 weeks' gestation, 3 months' postpartum and 6-months postpartum to assess baseline values and trial outcomes, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (12-25 weeks' gestation)
* subclinical and clinical levels of depression (Edinburgh Postnatal Depression Scale (EPDS) scores 8-16)
* ability to read and understand French.

Exclusion Criteria:

* EPDS score in the clinical range (≥ 17) or no symptoms (EPDS < 8)
* Positive screening of psychotic symptoms using the Psychosis Screening Questionnaire (PSQ)
* self-reported substance abuse problems.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 3 month postpartum depressive symptoms: The Edinburgh Perinatal/Postnatal Depression Scale (EPDS) | baseline (between gestational weeks 12-25) , 3 months postpartum
  The Edinburgh Perinatal/Postnatal Depression Scale (EPDS) assesses a score between 0 and 30. A score less than 8 means depression is unlikely. A score from 9 to 11 means depression is possible. A score from 12 to 13 means high possibility of depression. A score of 14 and higher means probable depression.

SECONDARY OUTCOMES:
Depressive symptoms: The Edinburgh Postnatal Depression Scale (EPDS) | 6 months postpartum
  The Edinburgh Perinatal/Postnatal Depression Scale (EPDS) assesses a score between 0 and 30. A score less than 8 means depression is unlikely. A score from 9 to 11 means depression is possible. A score from 12 to 13 means high possibility of depression. A score of 14 and higher means probable depression.
Change from baseline in Generalized Anxiety Disorder questionnaire (GAD-7) score | baseline (between gestational weeks 12-25) , 3 and 6 months postpartum
  Brief questionnaire about problems felt during the last 2 weeks, derived from the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) symptom criteria for GAD for a total score ranging from 0-21. Minimal (0-4), mild (5-9), moderate (10-14), and severe (15-21) severity ranges have been identified, with a clinical cutoff score of 8 indicating probable diagnosis of GAD
Anxiety related to pregnancy: Pregnancy-specific anxiety scale (PRAQ-R2) | baseline (between gestational weeks 12-25)
  The 10-item Pregnancy-specific anxiety scale revisited-2 (PRAQ-R2) by Van den Bergh to assess and identify pregnancy-specific anxiety in nulliparous women. Scores on each item are ranged from 1 (definitely not true) to 5 (definitely true). The items are divided into three subscales. The 1st subscale - Fear of giving birth, consists of three items. The 2nd subscale - Worries about bearing a physically or mentally handicapped child, consists of 4 items. The 3rd subscale -Concern about own appearance, consists of 3 items.
Stress: Perceived Stress Scale (PSS) | 6 months postpartum
  The Perceived Stress Scale is a 14-items questionnaire to measure the degree to which respondents find their lives unpredictable, uncontrollable and overloading. Individual scores on the PSS can range from 0 to 40, with higher scores indicating higher perceived stress.
Well-being: WHO-5 (World Health Organization) index | 3 months postpartum
  The 5-item WHO-5 well-being index is used to assess subjective psychological well-being.
Self-efficacy: General Self-Efficacy scale (GSE) | 3 months postpartum
  The 10-items General Self-Efficacy scale was created to assess a general sense of perceived self-efficacy with the aim in mind to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events.The minimum score is ten points and the maximum score is forty points for this scale.
Self-compassion: Self-Compassion Scale (SCS) | 3 months postpartum
  We used the corresponding items from the short SCS in the 26-item French questionnaire, to use a 10-item French questionnaire. For each item (e.g.; I'm kind to myself when I'm experiencing suffering), respondents are asked to indicate how often they behave in the stated manner. Each statement is rated on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always).
Sleep: Pittsburgh Sleep Quality Index (PSQI) | 3 months postpartum
  The Pittsburgh Sleep Quality Index (PSQI), a 19-items self-report questionnaire measuring sleep quality over a one-month interval.
Social Adjustment: Social Adjustment Scale - Self-report (SAS-SR) | 3 months postpartum
  The Screener version of the Social Adjustment Scale (SAS-SR) is a self-reported 14-item questionnaire derived from the Social Adjustment Scale interview. The questions measure expressive and instrumental performance over the past 2 weeks in six roles areas: work (paid or unpaid), social and leisure activities, relationships with extended family, role as marital partner, role as parent, and role within the family unit. Each area covers four expressive and instrumental categories: performance at expected tasks; the amount of friction with people; finer aspects of interpersonal relations; and feelings and satisfactions. Questions are rated on a five-point scale from which role area means and an overall mean can be obtained, with higher scores meaning greater impairment. The investigators used only the work subscale for this study
Marital satisfaction: Short Form of the Dyadic Adjustment Scale (DAS-7) | 3 months postpartum
  The 7-item Dyadic Adjustment Scale (DAS-7) is a shortened version of the original 32-item scale was created to assess multidimensional subjective satisfaction of marriage or similar dyads (93). In the shortened version, six items are rated on a six-point Likert-type scales (from "always agree" to "always disagree" or "all the time" to "never") and the seventh is rated on a seven-point scale (from "extremely unhappy" to "perfectly happy"). A 16-item version of the scale was translated in French and validated. We extracted the 7 items corresponding to DAS-7 from the 16-item French questionnaire.
Co-parenting: Co-parenting Relationship Scale (CRS) | 3 months postpartum
  The Co-parenting Relationship Scale multi-domain measure of the co-parenting relationship in dual parent families. The self-reported questionnaire contains 35 items and 7 subscales: Co-parenting Agreement, Co-parenting Closeness, Exposure, Conflict, Co-parenting Support, Co-parenting Undermining, Endorse Partner Parenting, and Division of Labor. Answers have a 7-point response scale ranging from "not true of us" to "very true of us"
Social support: Social Provisions | 6 months postpartum
  The initial 10-items Social Provisions Scale (SPS) was developed based on Weiss's model of social provisions. The model focus on five social need that can be fulfilled through relationships: guidance, reliable alliance, reassurance of worth, attachment and social integration. Each of the 5 subscales are represented by 2 positively worded statements and rated on a 4-point Likert scale from "1=strongly disagree" to "4=strongly agree"
Parenting practices: Parenting Cognitions and Behaviors Scale | 6 months postpartum
  The Parenting Cognitions and Behaviors Scale assesses parents' cognitions and behavioral tendencies that reflect the quality of their parental involvement with the infant. The scale has 32 items, measured on a Likert scale with scores ranging from 0 ("Not at all") to 10 ("Exactly"). The instrument has 6 dimensions: sense of parental efficacy, perceived impact of parenting, tendency to coerce, tendency to overprotect, parental affection, and parent's perception of the child's general qualities.
Change from 3 months post-partum at 6 month post partum child social, emotional and cognitive development: Ages and stages questionnaire 3rd edition (ASQ-3) | 3 and 6 months postpartum
  The Ages and Stages Questionnaire is a parent-reported scale designed to screen for developmental delays in children. The scale comprises 21 age-speciﬁc questionnaires, covering 1 through 66 months of age, each with six items in each of ﬁve developmental domains: communication, problem-solving, personal-social, gross motor, and ﬁne motor skills. Answers to each item are "yes," "sometimes," or "not yet", corresponding to scores of 10,5 and 0.
Child's temperament: Difficult Temperament Scale | 6 months postpartum
  The 7 items of the difficult temperament scale are taken from the Infant Characteristics Questionnaire (ICQ) of Bates, Freeland and Lounsbury, which is designed to measure the degree of difficulty a child presents to his or her parents. Parents are asked to indicate on a scale of 1 (easy) to 7 (difficult) how they perceive their baby's behavior when compared with that of an "average" or "typical" baby.
Personality disorders symptoms: Personality Inventory for DSM-5 Brief Form (PID-5 BF) | baseline (between gestational weeks 12-25)
  The brief form of the Personality Inventory for DSM-5 is a 25-item self-report questionnaire that measures the severity of the DSM-5-proposed personality pathology constructs of negative affectivity, detachment, antagonism, disinhibition, and psychoticism.
Gender roles: Bem Sex Role Inventory (BSRI) | 6 months postpartum
  The BEM Sex Role Inventory (BSRI) is a 30-items self-reported scale designed to evaluate gender. The items in the masculine subscale measure socially desirable masculine characteristics, with the central characteristic being "cognitive focus on getting the job done". The items in the feminine subscale are intended to measure socially desirable feminine characteristics, with the central characteristic being "affective concern for the welfare of others

OTHER OUTCOMES:
Health Service Utilization and Cost of Care Questionnaire | 6 months postpartum
  We reduced the questionnaire to 24 questions and translated it in French.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvana Côté, Principal Investigator — St. Justine's Hospital
Locations (1):
- St. Justine hospital, Montreal, Quebec, Canada

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT05110456/Prot_SAP_000.pdf